CLINICAL TRIAL: NCT04831060
Title: Characterization of the Immuno-inflammatory Response Involved in Bone Destruction During Periodontitis: Study With Biological Collection
Brief Title: Periodontitis and Inflammation
Acronym: CB-PARO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200784
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Peri-Implantitis
Keywords: Periodontitis; Inflammation; Cytokines; Diabetes Mellitus; peri-implantitis
MeSH Terms: conditions — Periodontitis; Peri-Implantitis; Inflammation; Diabetes Mellitus | interventions — Tooth Exfoliation; Periodontal Debridement; Gingivectomy; Crown Lengthening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial, gum fluid and saliva collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case Periodontitis: Patients with stage 3 or 4 periodontitis
  Interventions: Procedure: Periodontal or peri-implantitis treatment
- Case peri-implantitis: Patients should present at least 1 implant with peri-implantitis
  Interventions: Procedure: Periodontal or peri-implantitis treatment
- Control (healthy periodontium): Patients with gingival health on intact or reduced periodontium without a history of periodontitis or peri-implantitis and requiring surgical care such as dental avulsion or pre-prosthetic periodontal surgeries or aesthetic surgeries
  Interventions: Procedure: Control treatment

INTERVENTIONS:
Procedure: Periodontal or peri-implantitis treatment — For Cases :
  * Inclusion; Bacterial sampling, gingival fluid and unstimulated saliva collection; Teaching of oral hygiene techniques.
  * Non-surgical periodontal or peri-implantal treatment
  * At 3 months = periodontal or peri-implantal reevaluation; Bacterial sampling, gingival fluid and unstimulated saliva collection
  * If periodontal or peri-implantal pockets greater than 5mm and bleeding persist: surgery and gingival explant sampling
  * At 3 months post-surgery = periodontal or peri-implantal re-evaluation; Bacterial sampling, gingival fluid and unstimulated saliva collection
  * Maintenance
  Other Names: Scaling and root planning; periodontal debridement; periodontal or peri-implantal surgery; open flap debridement; gingivectomy; crown lengthening; periodontal plastic surgery; pre-prosthetic periodontal surgery
  Groups: Case Periodontitis; Case peri-implantitis
Procedure: Control treatment — For Controls:
  * Inclusion; Bacterial sampling, gingival fluid and unstimulated saliva collection, teaching of oral hygiene techniques.
  * Plastic or pre-prosthetic surgery = gingival explant sampling
  * Healing control at 15 days
  Groups: Control (healthy periodontium)

SUMMARY:
Today, to understand pathogenic mechanisms involved in periodontitis and peri-implantitis remains a challenge to identify biomarkers or therapeutic targets to improve prevention and screening, as well as the effectiveness of periodontitis and peri-implantitis treatments. The aim is to characterize, in vivo, specific molecular markers reflecting the activity of the pathology, which could lead to

* improve the knowledge of the pathogenesis of periodontitis and peri-implantitis;
* determine target molecules involved in tissue destruction;
* determine molecular profiles of patients at local and systemic risk;
* determine therapeutic targets

For this purpose, biological samples will be collected (plaque, saliva, crevicular fluid) from patients with periodontitis or peri-implantitis stage 3 or 4 versus patients with a healthy periodontium. Biological samples will be collected before and all along the periodontal or peri-implantal treatment. Gingiva explants collection will be sampling within the surgical procedures (if they are needed).

The primary objective is to investigate tissue and cellular expression of molecular markers associated with periodontal destruction during periodontitis or peri-implantitis in relation to periodontal infection and systemic changes in host response. A characterization of the cytokines in gingival fluid and unstimulated saliva (Luminex® technique) of patients with periodontitis or peri-implantitis versus without periodontitis or peri-implantitis will be done.

The secondary objective is to study the influence of periodontitis on systemic pathologies via serum analysis of molecules and bacteria involved in periodontal destruction. Immunofluorescence evaluation of protein expression and distribution (inflammatory mediators, inflammatory pathway signaling proteins) in gingival explants, characterization of proteases (MMP) present in gingival fluid and unstimulated saliva (Luminex® technique) and microbiological analysis of the subgingival biofilm (by quantitative PCR).

DETAILED DESCRIPTION:
Today, to understand pathogenic mechanisms involved in periodontitis and peri-implantitis remains a challenge to identify biomarkers or therapeutic targets to improve prevention and screening, as well as the effectiveness of periodontitis and peri-implantitis treatments. The aim is to characterize, in vivo, specific molecular markers reflecting the activity of the pathology, which could lead to

* improve the knowledge of the pathogenesis of periodontitis and peri-implantitis;
* determine target molecules involved in tissue destruction;
* determine molecular profiles of patients at local and systemic risk;
* determine therapeutic targets

The research focuses on the characterization of the immuno-inflammatory response involved in periodontitis and peri-implantitis. A characterization of the mediators or cells involved will be performed from biological samples (gingival fluid, unstimulated saliva, gingival explants). The gingival fluid is composed of serum inflammatory exudate and inflammatory mediators produced locally in the periodontal pocket. Unstimulated saliva is a biological fluid composed in part of the gingival fluid that drains into it. It has the advantage of being easier to collect (larger quantity, collection by any health professional).

This is a non-interventional, cross-sectional, multicenter, prospective, open-label, non-randomized study to collect tissue, crevicular, salivary, and serum samples as part of the patient's routine care in oral medicine departments to form a biological collection. The samples and the clinical data of the patients (excel file with anonymized data and locked by a password) will be transferred to UMR1333 for their analysis.

Patients will be recruited in the oral medicine departments of AP-HP hospitals (Charles Foix (Ivry/seine) and Rothschild (Paris) by periodontists in three groups (cases = periodontitis or peri-implantitis and controls = healthy periodontium but patients requiring surgical care).

The time-line of the research is consistent with the usual patient management in oral medicine departments. Inclusion period is 60 months. There is no specific follow-up due to the research.

Gingival tissue sampling during surgery of patients will be performed after their inclusion.

ELIGIBILITY:
Inclusion Criteria:

Common criteria for all patient groups

* Patient > 18 years old
* Patient affiliated to a social security system, beneficiary or beneficiary of a right other than AME
* Patient who speaks and understands French well enough to be able to read and understand the study information note.
* Patient who does not object to his participation in the study

Specific criteria:

- Case Periodontitis: Patient with localized or generalized periodontitis, stage 3 or 4. The diagnosis of periodontitis is based on the elements found during the interview and clinical examination

- Case peri-implantitis: Patients with at least 1 implant affected by peri-implantitis. Diagnosis is based on the findings of the interview, clinical examination and radiographic examination.

Control group:

Patient with gingival health on intact or reduced periodontium with no history of periodontitis or peri-implantitis and requiring surgical care such as dental avulsion and pre-prosthetic periodontal corrective/aesthetic surgeries (coronal elongation, neck alignment.)

Exclusion Criteria:

* Patients who have received antibiotic prophylaxis, antibiotic therapy, or anti-inflammatory treatment within 3 months prior to inclusion
* Pregnant or breastfeeding women
* Patient included in another interventional research protocol or in a period of exclusion.
* Patients under guardianship, curatorship or legal protection.
* Patient having expressed his opposition to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study concerns adult patients consulting the oral medicine departments of Hôpital Charles Foix (AP-HP, Ivry sur Seine) and Hôpital Rothschild (AP-HP, Paris) - Patients:
  Patients should have:
  - localized or generalized periodontitis of stage 3 or 4. The diagnosis of periodontitis is based on the elements noted during the interview and the clinical examination.
  Or
  * at least 1 implant with peri-implantitis. The diagnosis is based on the findings of the interview, clinical examination and radiographic examination.
  * Controls:
  Patients with gingival health on intact or reduced periodontium with no history of periodontitis and requiring surgical care such as dental avulsion and pre-prosthetic periodontal corrective/aesthetic surgeries (coronal elongation, neck alignment
Sampling Method: Non-Probability Sample
Enrollment: 219 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Characterization of a panel of cytokines in gingival fluid of patients with periodontitis versus without periodontitis | 1 month once the collection is completed
  Analysis of gingival fluids and unstimulated saliva by the Luminex allows detection and quantification of 15 cytokines (IL- 1α, IL- 1β, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-15, IL-17, IL-18, IFN γ, TNF) simultaneously

SECONDARY OUTCOMES:
Cytokines expression in periodontal cells | 6 months once the collection is completed
  Analysis of cytokines, inflammation pathways and inflammation cells by histological analysis (immunofluorescence) of surgical specimens.
Cytokines expression in periodontal cells | 6 months once the collection is completed
  Immunofluorescence evaluation of protein distribution (inflammatory mediators, inflammatory pathway signaling proteins) in gingival explants (confocal microscopy analysis).
Microbiological analysis of the subgingival biofilm determination of the percentage of periodontopathogens. | 3 months once the collection is completed
  assessment through RT-PCR
Characterization of proteases (MMP) present in gingival fluid and unstimulated saliva | 1 month once the collection is completed
  assessment through Luminex®

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service d'odontologie, hôpital Charles Foix, Ivry-sur-Seine
  - Dentistry department- Rothschild hospital, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.